CLINICAL TRIAL: NCT01342445
Title: Effects of Vyvanse on the Behavioral, Academic, and Psychosocial Functioning of College Students With ADHD
Brief Title: Effects of LDX on Functioning of College Students With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Lehigh University (Other)
Responsible Party: Principal Investigator, Lisa Weyandt, Professor, University of Rhode Island
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Shire-80000311112
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- lisdexamfetamine dimesylate (Experimental): All participants will be assessed across five conditions (baseline, placebo, 30-mg, 50-mg, & 70-mg) in a double-blind, crossover design
  Interventions: Drug: lisdexamfetamine dimesylate; Drug: Placebo

INTERVENTIONS:
Drug: lisdexamfetamine dimesylate — 30-mg, 50-mg, 70-mg administered for one week in context of double-blind, placebo-controlled crossover design
  Other Names: Vyvanse; LDX
Drug: Placebo

SUMMARY:
The purpose of this study was to evaluate the effects of lisdexamfetamine dimesylate, a prodrug stimulant, on the behavioral, academic, and psychosocial functioning of college students with attention-deficit/hyperactivity disorder (ADHD). Twenty-five college students with ADHD from two universities (University of Rhode Island and Lehigh University) completed a within-subject, placebo-controlled research trial. Dependent measures tapping behavioral, psychosocial, and academic functioning were completed on a weekly basis across five conditions (baseline, placebo, and 30-mg, 50-mg, and 70-mg lisdexamfetamine).

DETAILED DESCRIPTION:
Objective: Evaluate stimulant medication on symptoms and functioning for college students with ADHD using double-blind, placebo-controlled, crossover design. Method: Participants included 24 college students with ADHD and 26 college students without psychopathology. Lisdexamfetamine dimesylate (LDX) examined for ADHD participants over five weekly phases (no-drug baseline, placebo, 30, 50, & 70-mg LDX per day). Self-report rating scales of functioning and direct assessment of ADHD symptoms, verbal learning/memory, and adverse side-effects were collected (baseline only for control students).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Statistical Manual of Mental Disorders 4th edition-text revision (DSM-IV-TR) criteria for ADHD based on self- and parent-report using questionnaires and clinical interview

Exclusion Criteria:

* significant cardiac condition based on medical history and/or physical examination
* significant substance abuse based on self-report and toxicology screen at intake
* significant symptoms of major depressive disorder, bipolar disorder, or thought disorder based on initial diagnostic interview

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Weyandt, PhD, Principal Investigator — University of Rhode Island
Locations (2):
- United States (2):
  - Department of Education and Human Services, Lehigh University, Bethlehem, Pennsylvania
  - Department of Psychology, University of Rhode Island, Kingston, Rhode Island

REFERENCES:
- [Result] Dupaul GJ, Weyandt LL, Rossi JS, Vilardo BA, O'Dell SM, Carson KM, Verdi G, Swentosky A. Double-blind, placebo-controlled, crossover study of the efficacy and safety of lisdexamfetamine dimesylate in college students with ADHD. J Atten Disord. 2012 Apr;16(3):202-20. doi: 10.1177/1087054711427299. Epub 2011 Dec 12. PMID 22166471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from student disabilities and health service offices at two univer- sities in the Northeastern United States (one public and one private).
Pre-assignment Details: Almost all participants completed all stages of the trial. One participant withdrew from the study after a possible adverse reaction.
Groups:
- Healthy Controls: All participants completed the Conners' Adult ADHD Rating Scales-Short Form (CAARS) and Behavior Rating Inventory of Executive Functioning-Adult Version (BRIEF) at baseline only and received no drug.
- Attention-deficit/Hyperactivity Disorder (ADHD) Participants: All participants completed the Conners' Adult ADHD Rating Scales-Short Form (CAARS) and Behavior Rating Inventory of Executive Functioning-Adult Version (BRIEF) at baseline and were randomly assigned to one of six medication orders using placebo, 30-mg, 50 and 70 mg lisdexamfetamine dimesylate (LDX) in the context of a double-blind, crossover design, with repeated measures at the end of each drug phase. Phase orders (following baseline) were assigned in a counterbalanced fashion across participants. To avoid starting any participant with the highest dosage, the 50-mg condition always preceded the 70-mg condition. Each phase was conducted for 1 week, and therefore, the total trial took place over 5 weeks and was able to be completed during a single semester. Participants ingested one pill per day on awakening.
Period: Overall Study
Arm/Group | Healthy Controls | Attention-deficit/Hyperactivity Disorder (ADHD) Participants
Started | 26 | 24
Completed | 26 | 22
Not Completed | 0 | 2
Not completed — Experienced side effects | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- ADHD Participants: All participants completed the Conners' Adult ADHD Rating Scales-Short Form (CAARS) and Behavior Rating Inventory of Executive Functioning-Adult Version (BRIEF) at baseline and were randomly assigned to one of six medication orders using placebo, 30-mg, 50 and 70 mg LDX in the context of a double-blind, crossover design, with repeated measures at the end of each drug phase. Phase orders (following baseline) were assigned in a counterbalanced fashion across participants. To avoid starting any participant with the highest dosage, the 50-mg condition always preceded the 70-mg condition.
- Total: Total of all reporting groups
Arm/Group | ADHD Participants | Healthy Controls | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.17 (1.2) | 20 (1.1) | 20.17 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: participants] — Not all ethnicity categories are covered, and a participant may be counted in more than one ethnicity
  participants
    White non-Hispanic | 22 | 21 | 43
    African American | 1 | 0 | 1
    Hispanic | 0 | 3 | 3
    Asian/Pacific Islander | 1 | 1 | 2
    Indian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
Conners Adult Rating Scale [Mean (Standard Deviation); unit: T score] — The Conners was converted to a T score with a mean of 50 and standard deviation of 10. Higher scores represent more severe ADHD symptoms.
  T score | 58.04 (7.51) | 36.12 (4.98) | 47.08 (NA) — The standard deviation was not pre-specified to be calculated.
BRIEF [Mean (Standard Deviation); unit: T score] — The BRIEF was converted to a T score with a mean of 50 and a standard deviation of 10. Higher scores represent poorer levels of functioning.
  T score | 65.41 (11.661) | 44.31 (7.62) | 54.86 (NA) — The standard deviation was not prespecified to be calculated for the total sample.
Year in College [Number; unit: participants]
  Freshman | 3 | 5 | 8
  Sophomore | 7 | 6 | 13
  Junior | 4 | 7 | 11
  Senior | 10 | 8 | 18
Father's level of education [Number; unit: participants]
  Less than high school (HS) | 0 | 0 | 0
  HS diploma or equivalent | 6 | 6 | 12
  Some college | 2 | 3 | 5
  Bachelor's degree | 11 | 7 | 18
  Graduate degree | 5 | 9 | 14
  Training program or certificate | 0 | 1 | 1
Mother's level of education [Number; unit: participants]
  Less than high school (HS) | 1 | 0 | 1
  HS diploma or equivalent | 3 | 3 | 6
  Some college | 5 | 4 | 9
  Bachelor's degree | 9 | 8 | 17
  Graduate degree | 6 | 9 | 15
  Training program or certificate | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Conners Adult ADHD Rating Scale - Short Version (CAARS)
Description: CAARS ADHD Index, adult self-report measure of ADHD symptoms. T-scores (mean = 50; standard deviation = 10) for all subscales on the short version were used as dependent measures with higher scores representing greater ADHD symptomatology (and ultimately a worse outcome in this study).
Time Frame: after receiving Placebo or LDX for 1 week
Measure: Mean (Standard Deviation); unit: T score
Groups:
- Placebo: All participants receiving Placebo for 1 week in a double-blind, crossover design
- LDX 30-mg: All participants receiving 30-mg LDX for 1 week in a double-blind, crossover design
- LDX 50-mg: All participants receiving 50-mg LDX for 1 week in a double-blind, crossover design
- LDX 70-mg: All participants receiving 70-mg LDX for 1 week in a double-blind, crossover design
Arm/Group | Placebo | LDX 30-mg | LDX 50-mg | LDX 70-mg
Number analyzed (Participants) | 22 | 22 | 22 | 22
T score | 50.59 (10.975) | 46.86 (9.939) | 47.32 (10.092) | 45.36 (10.790)
Statistical Analysis 1: Comparison: Placebo vs LDX 30-mg vs LDX 50-mg vs LDX 70-mg; This was a within-subject crossover design with all participants going through a no-drug baseline followed by placebo and three dosages of LDX, with the latter four conditions in a randomly assigned, counterbalanced order. The comparison condition was the placebo condition; Test type: Superiority or Other; p < 0.001, ANOVA — we adjusted p values to control for the false discovery rate using procedures described by Benjamini and Hochberg (1995). Thus, an alpha value of .021 was used as significance threshold; F(4, 84) = 10.9 This was a one-way ANOVA with repeated measures across dosage conditions (no drug baseline, placebo, 30-mg, 50-mg, 70-mg LDX); Partial eta squared = .34

2. Primary Outcome: Behavior Rating Inventory of Executive Function - Adult (BRIEF-A)
Description: BRIEF-A is a standardized self-report measure that captures adults' views of their own self-regulation in their everyday environment. Metacognition Index T-scores (mean = 50; standard deviation = 10) were used as dependent measures with higher scores representing greater deficit in planning/organizational skills critical for college success.
Time Frame: after receiving Placebo or LDX for 1 week
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Placebo | LDX 30-mg | LDX 50-mg | LDX 70-mg
Number analyzed (Participants) | 22 | 22 | 22 | 22
T score | 65.91 (13.023) | 59.23 (14.088) | 57.64 (14.012) | 54.91 (13.219)
Statistical Analysis 1: Comparison: Placebo vs LDX 30-mg vs LDX 50-mg vs LDX 70-mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .001, ANOVA — [p-value comment as in outcome 1, analysis 1]; F(4, 84) = 8.14 This was a one-way ANOVA with repeated measures across dosage conditions (no drug baseline, placebo, 30-mg, 50-mg, 70-mg LDX); partial eta squared = 0.28

ADVERSE EVENTS:
Time Frame: Adverse event data was collected and updated on a daily basis during the 1 week receiving placebo or LDX.
Description: If an adverse event occurred, the prescribing nurse would review with the participant and review risks. Adverse Events were only collected for the 24 participants who actually met inclusion criteria for ADHD and thus qualified for the medication trial
Arm/Group | Placebo | LDX 30-mg | LDX 50-mg | LDX 70-mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 2/24 | 0/24 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | LDX 30-mg (N=24) | LDX 50-mg (N=24) | LDX 70-mg (N=24)
Possible Heart Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — This was the adverse event for both participants. This occurred during week 1 of the medication trial in which both participants were taking an active dosage of 30mg.

LIMITATIONS AND CAVEATS:
No notable limitations or caveats are noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No